CLINICAL TRIAL: NCT05035108
Title: A Clinical Study of hiHep Cells for Bioartificial Liver After Extensive Hepatectomy
Brief Title: The Treatment of Bioartificial Liver With hiHep Cells After Extensive Hepatectomy
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sir Run Run Shaw Hospital (Other)
Collaborators: Hexaell Biotech Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Xiujun Cai, The director of Sir Run Run Shaw Hospital, Sir Run Run Shaw Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SRRSH20201110-8
Record Dates: First submitted 2021-05-31; First posted 2021-09-05 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Hepatoma Resectable

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- extensive hepatectomy patient (Experimental): hiHep bioartificial liver therapy
  Interventions: Biological: hiHep bioartificial liver therapy

INTERVENTIONS:
Biological: hiHep bioartificial liver therapy — HiHep cell bioartificial liver treatment was performed 48-72 hours after extensive hepatectomy. Temporary hemodialysis tube for large vein (jugular vein or femoral vein) is indwelled before treatment. Before treatment, prepare hiHeps-BAL in a biological safety cabinet that meets clinical standards, connect the corresponding tubing to the Jianfan DX-10 blood purification machine, and prefill with heparin saline. Half an hour before treatment, the patient was pre-heparinized (heparin about 600iu) and dexamethasone to prevent allergic reactions. The patient enters the ICU, the monitor is connected to the corresponding pipeline, the arterial pump 120-160ml/min, the slurry pump 30-40ml/min, the circulating pump 75-100ml/min, the duration is 4-6h.

SUMMARY:
It is a prospective, non-randomized, single-arm cohort study. A total of 10 patients will be included in this study. Based on standardized treatment, the treatment of bioartificial liver device will be applied 48-72 hours after extensive hepatectomy. The bioartificial liver device consists of clinical-grade human-induced hepatocytes (hiHep) generated from human fibroblasts via transdifferentiation. In order to evaluate the security and effectiveness of the device, liver function, liver volume, the incidence of liver failure and other results will be analyzed.

DETAILED DESCRIPTION:
Include large-scale hepatectomy patients who meet the Inclusion criteria into the experimental group. Patient will be sent to ICU monitoring after surgery , the investigators will evaluate the blood routine, liver and kidney function, blood coagulation function, and immune inflammation indicators on the first day after surgery, and large veins will be temporarily indwelled within 48-72 hours Hemodialysis tube, then take artificial liver treatment which lasts 4-6h, follow-up test results on the 1st day, 3rd day, 7th day, 1 month and 3 months about blood routine, liver and kidney function, coagulation function, blood ammonia, Immune inflammation indicators, imaging examinations (CT or MR) at 7 days, 1 month and 3 months after treatment, to evaluate the recovery of liver function and liver regeneration after artificial liver treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed as liver cancer, hepatolithiasis, benign liver tumor, with clear indications for liver resection;
2. Liver function Child A-B;
3. There is no contraindication to surgery for cardiopulmonary function;
4. The expected remaining liver volume/standard liver volume is less than 50%;

Exclusion Criteria:

1. In the late stage of the disease, patients with frequent symptoms such as cerebral edema accompanied by cerebral herniation and clinical evidence indicating intracranial hemorrhage;
2. PaO2/FiO2 is less than 200 and cannot be corrected;
3. Patients with diffuse intravascular coagulation;
4. Those with active bleeding;
5. Uncontrolled infection;
6. The platelet count is less than 50,000/μL and cannot be corrected;
7. There is no blood vessel available for dialysis treatment;
8. HIV, HDV or HCV positive;
9. Drug abuse within 1 year;
10. Those with severe systemic circulatory failure;
11. Those who are highly allergic to the drugs used in the treatment process, such as plasma, heparin, protamine, etc.;
12. Combined pregnancy;
13. Patients with hepatorenal syndrome;
14. Patients with autoimmune liver disease;
15. Patients with non-alcoholic fatty liver and hereditary liver diseases (Wilson syndrome and a-antitrypsin deficiency);
16. Other conditions that the clinician believes cannot tolerate the treatment.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-09-05 (Actual); Primary Completion 2030-11-30 (Estimated); Study Completion 2030-11-30 (Estimated)

PRIMARY OUTCOMES:
The incidence of adverse events (safety and tolerability). | 3 months after therapy
  Record adverse events (AE), serious adverse events (SAE), and AEs (TEAE) that occurred during treatment.

SECONDARY OUTCOMES:
Patient's recovery of liver function | 1day,3day,7day,1month,3 months after therapy
  Through child-pugh liver function grading standard and changes in ALT, AST, AKP, r-GGT, TBil, DBil, ALB to evaluate liver function.
Rate of liver proliferation | 7day,1month,3 months after therapy
  Remaining liver growth rate (calculation of residual liver volume based on CT three-dimensional reconstruction).
Incidence of liver failure | 1day,3day,7day,1month,3 months after therapy
  Use Guidelines for The Diagnosis and Treatment of Liver Failure (exclude liver failure caused by surgical hemodynamic problems).
Complication rate | 1day,3day,7day,1month,3 months after therapy
  Such as pleural effusion, hydrops abdominis, hemorrhage, bile leakage.
Immunoinflammatory index | 1day,3day,7day,1month,3 months after therapy
  Changes in PCT, hCRP, immune globulin (IgA, IgM, IgG), complement (C3, C4) after the treatment.
Renal function | 1day,3day,7day,1month,3 months after therapy
  Record the changes in creatinine and urea nitrogen, calculate GFR through MDRD or CKD-EPI formula to evaluate renal function by classification standards for renal insufficiency.
Electrolyte level | 1day,3day,7day,1month,3 months after therapy
  Changes in the concentration of Na+, K+, Cl+, Ca+ in blood before and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Yifan Wang, MD, Principal Investigator — Sir Run Run Shaw Hospital
Locations (1):
- Department of General Surgery, Institute of Minimally Invasive Surgery, Sir Run Run Shaw Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No